CLINICAL TRIAL: NCT02593331
Title: A Phase Ia, Randomized, Blinded, Placebo-Controlled, Ascending Single Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Subcutaneous and Intravenous BFKB8488A in Otherwise Healthy Overweight and Obese Volunteers With Likely Insulin Resistance
Brief Title: Study to Evaluate Safety, Tolerability, and Pharmacokinetics of BFKB8488A in Otherwise Healthy Overweight and Obese Participants With Likely Insulin Resistance
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GC29819
Record Dates: First submitted 2015-10-20; First posted 2015-11-02 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Placebo (Placebo Comparator): Participants will receive placebo matching to BFKB8488A.
  Interventions: Other: Placebo
- BFKB8488A SC (Experimental): Participants will receive single ascending SC dose of BFKB8488A in each dose escalation cohort.
  Interventions: Drug: BFKB8488A
- BFKB8488A IV (Experimental): Participants will receive single IV dose of BFKB8488A.
  Interventions: Drug: BFKB8488A

INTERVENTIONS:
Drug: BFKB8488A — Participants will receive either a single escalated dose of BFKB8488A administered SC or a single dose of BFKB8488A administered IV on Day 1.
  Arms: BFKB8488A IV; BFKB8488A SC
Other: Placebo — Participants will receive a single dose of placebo on Day 1.
  Arms: Placebo

SUMMARY:
This study will evaluate the safety and tolerability profile of BFKB8488A following subcutaneous (SC) administration in overweight and obese participants (body mass index [BMI] greater than [>] 27 to less than or equal to [</=] 40 kilograms per square meter [kg/m^2]) with markers of insulin resistance. Single ascending fixed doses of BFKB8488A will be evaluated. Participants will be randomized into 7 sequential ascending fixed-dose cohorts of BFKB8488A SC or placebo and safety reviews will be performed before escalation to higher dose cohorts. Additionally, following the ascending fixed-dose SC cohorts, a separate cohort will open to evaluate the PK of BFKB8488A after intravenous (IV) administration.

ELIGIBILITY:
Inclusion Criteria:

* Participants with BMI >/=30 kg/m^2 and </=40 kg/m^2 or BMI >27 kg/m^2 and <30 kg/m^2 and Homeostatic Model Assessment-Insulin Resistance (HOMA-IR) >3.60 or waist circumference >100 centimeters (cm) (males) or 88 cm (females) or fasting plasma insulin >/=15 milli international unit per liter (mIU/L) or fasting plasma glucose >/=100 milligrams per deciliter (mg/dL) and <126 mg/dL or hemoglobin A1c (HbA1c) >5.6 percent (%) and <6.5%
* Negative pregnancy test

Exclusion Criteria:

* A diagnosis of Type 2 diabetes mellitus at any time
* Pregnant, lactating or intending to become pregnant during the study or within 3 months after the study dose is administered
* Uncontrolled intercurrent illness or any psychiatric illness
* Participants actively involved in a weight loss or dietary program within the last 6 months
* History of surgical procedures for weight loss
* History of eating disorder
* Uncontrolled hypertension (systolic >/=140 millimeter of mercury [mmHg] or diastolic blood pressure >/=90 mmHg) either on or off therapy at screening or Day -2
* Fasting triglycerides >500 mg/dL (5.64 millimoles per liter [mmol/L]) or low density lipoprotein (LDL) >160 mg/dL (4.14 mmol/L) at screening
* Any serious medical condition or abnormality in clinical laboratory tests

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2015-10-29 (Actual); Primary Completion 2017-03-28 (Actual); Study Completion 2017-03-28 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events | From baseline up to 20 Weeks

SECONDARY OUTCOMES:
Serum BFKB8488A Concentration | SC Cohort: predose (Hour 0), 4, 24, 72 hours post Day 1 dose, Days 6, 8, 11, 15, 22, 29, 36, 43, 57, 85, 113; IV Cohort: end of infusion on Day 1, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72 hours post Day 1 dose, Days 6, 8, 15, 22, 29, 36, 43

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Profil Institute for Clinical Research Inc., Chula Vista, California, United States